CLINICAL TRIAL: NCT07325370
Title: Right Dorsolateral Prefrontal Cortex-Targeted fNIRS-BCI Closed-loop Neurofeedback for Anxiety Relief and Cardiac Autonomic Regulation in Women With Recurrent Pregnancy Loss: a Randomized, Sham-controlled Clinical Trial
Brief Title: Cardiac Autonomic and Anxiety Regulation Via Closed-loop nEurofeedback in Recurrent Pregnancy Loss
Acronym: CARE-RPL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Medical College (Other)
Collaborators: Central Hospital Affiliated to Shenyang Medical Collage (Other)
Responsible Party: Principal Investigator, Lin Tao, Assoc.Prof., Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARE-RPL
Record Dates: First submitted 2025-12-22; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Pregnancy Loss; Anxiety
Keywords: Recurrent pregnancy loss; Anxiety disorders; Right dorsolateral prefrontal cortex; Functional near-infrared spectroscopy; Brain-computer interface; Closed-loop neurofeedback; Cardiac autonomic function; Brain-heart coupling
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, parallel-group, two-arm interventional study model with 1:1 allocation. Eligible women with recurrent pregnancy loss and comorbid anxiety will be assigned to real right DLPFC fNIRS-BCI online closed-loop neurofeedback or sham feedback. Both arms will use an identical training schedule and procedures: a 3-day adaptation phase followed by 3 weeks of formal training (15 sessions; one weekday session/day; ~20 min/session) using a block design (20 blocks/session; 60 s per block: 20 s rest + 40 s slow-wave acoustic cueing with a 1 Hz amplitude-modulated tone). fNIRS will be recorded in all sessions; ECG will be recorded only in session 1 for HR/HRV mechanistic outcomes. Outcomes will be assessed at baseline, end of treatment, and 3-month follow-up.
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking (blinding) will be implemented at multiple levels. Participants will be blinded to group assignment, and both groups will receive identical slow-wave acoustic cueing, session structure, instructions, and an indistinguishable on-screen feedback interface with the numerical threshold concealed. Outcome assessors (clinical raters) and data analysts/statisticians will remain blinded throughout data collection and primary analyses. Only the session operator responsible for loading group-specific neurofeedback parameters will be unblinded, and will not participate in outcome assessments or statistical analyses. Emergency unblinding will be permitted only when clinically necessary for participant safety and will be documented according to prespecified procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a real-feedback intervention group (Active Comparator): Participants will receive right DLPFC targeted fNIRS-BCI online closed-loop neurofeedback delivered with slow-wave acoustic cueing. Training includes a 3-day adaptation phase followed by 3 weeks of formal training (15 weekday visits; about 20 minutes per visit) using a block design (20 blocks per visit; 60 seconds per block: 20 seconds rest + 40 seconds slow-wave acoustic cueing with a 1 Hz sinusoidally amplitude-modulated pure tone at about 60 dB). During each cueing period, real-time right DLPFC activation estimated from fNIRS is displayed as a visual activation bar; participants apply volitional strategies to downregulate activity below a concealed threshold line (T = -3.3; approximating p = 0.001). fNIRS is recorded in all visits; ECG is recorded on the first formal training day only for HR/HRV measures.
  Interventions: Device: Right DLPFC fNIRS-BCI closed-loop neurofeedback (real feedback)
- a sham-feedback control group (Sham Comparator): Participants will receive sham fNIRS-BCI neurofeedback targeting the right DLPFC under procedures identical in appearance and schedule to the real-feedback arm, including the same slow-wave acoustic cueing and block design (20 blocks per visit; 60 seconds per block: 20 seconds rest + 40 seconds cueing with a 1 Hz sinusoidally amplitude-modulated pure tone at about 60 dB). fNIRS is recorded in all visits; ECG is recorded on the first formal training day only for HR/HRV measures. The on-screen interface and concealed threshold line are identical; however, feedback parameters are configured to substantially weaken effective coupling between the displayed activation bar and the participant's instantaneous neural activity (T = -1; approximating p = 0.31), making stable volitional control unlikely while preserving blinding.
  Interventions: Device: Right DLPFC fNIRS-BCI neurofeedback (sham feedback)

INTERVENTIONS:
Device: Right DLPFC fNIRS-BCI closed-loop neurofeedback (real feedback) — This device-based intervention delivers fNIRS-BCI online closed-loop neurofeedback targeting the right dorsolateral prefrontal cortex (right DLPFC) with slow-wave acoustic cueing. Participants complete a 3-day adaptation phase followed by 3 weeks of formal training (15 weekday visits; about 20 minutes per visit). Each visit includes 20 blocks (60 seconds per block: 20 seconds rest + 40 seconds slow-wave acoustic cueing with a ~60 dB, 1 Hz sinusoidally amplitude-modulated pure tone). During each cueing period, real-time right DLPFC HbO activity estimated from fNIRS is displayed as a visual activation bar, and participants apply volitional strategies to downregulate activity below a concealed threshold line (T = -3.3; approximating p = 0.001). fNIRS is recorded in all visits; ECG is recorded on the first formal training day only for HR/HRV mechanistic measures.
  Arms: a real-feedback intervention group
Device: Right DLPFC fNIRS-BCI neurofeedback (sham feedback) — This device-based sham intervention uses the same fNIRS-BCI neurofeedback interface, slow-wave acoustic cueing, and training schedule as the real-feedback arm. Participants complete a 3-day adaptation phase followed by 3 weeks of formal training (15 weekday visits; about 20 minutes per visit) using 20 blocks per visit (60 seconds per block: 20 seconds rest + 40 seconds slow-wave acoustic cueing with a ~60 dB, 1 Hz sinusoidally amplitude-modulated pure tone). fNIRS is recorded in all visits; ECG is recorded on the first formal training day only for HR/HRV measures. The displayed activation bar and concealed threshold line are configured to substantially weaken effective coupling to the participant's instantaneous neural activity (threshold setting: T = -1; approximating p = 0.31), making reliable volitional control unlikely while preserving blinding.
  Arms: a sham-feedback control group

SUMMARY:
The goal of this clinical trial is to learn whether right dorsolateral prefrontal cortex (right DLPFC)-targeted fNIRS-BCI online closed-loop neurofeedback, delivered with slow-wave acoustic cueing, can reduce anxiety symptoms and improve cardiac autonomic regulation in women with recurrent pregnancy loss (RPL) and comorbid anxiety (women aged 18-45 years, right-handed, currently not pregnant or in a missed miscarriage state).

The main questions it aims to answer are:

Does real neurofeedback increase the proportion of participants who achieve an anxiety treatment response (defined as ≥50% reduction in Hamilton Anxiety Rating Scale [HAMA] total score from baseline) compared with sham feedback, at end of treatment and at 3-month follow-up? Is the intervention safe and well tolerated, as reflected by between-group differences in adverse events during the training period? Do brain and autonomic measures show between-group differences during the first formal session, including right DLPFC HbO downregulation, interhemispheric DLPFC synchronisation, heart rate (HR), and heart rate variability (HRV) indices? Researchers will compare real right DLPFC neurofeedback to sham feedback (identical procedures and displays but weakened coupling to real-time neural activity) to see if real neurofeedback improves anxiety outcomes and brain-heart autonomic regulation.

Participants will:

Complete screening, baseline clinical assessments, and physical examination Be randomly assigned (1:1) to real neurofeedback or sham feedback Complete 3 days of adaptation training followed by 3 weeks of training (15 sessions; one weekday session per day; ~20 minutes each) using a block design with slow-wave acoustic cueing (1 Hz amplitude-modulated tone; 20 s rest + 40 s cueing per block; 20 blocks/session) Undergo fNIRS recording in all sessions, with ECG recorded in session 1 only (for HR/HRV analyses) Receive matched, guideline-informed cognitive-behavioural therapy (CBT) during the intervention period Complete anxiety-related assessments at baseline, ~1 hour after the final session, and 3 months after treatment, with adverse events monitored throughout the intervention period

DETAILED DESCRIPTION:
This study is a mechanistically informed, prospective, randomized, sham-controlled, parallel-group clinical trial designed to evaluate whether right dorsolateral prefrontal cortex (right DLPFC)-targeted fNIRS-BCI online closed-loop neurofeedback, delivered with slow-wave acoustic cueing, improves anxiety symptoms and cardiac autonomic regulation in women with recurrent pregnancy loss (RPL) and comorbid anxiety. Participants who meet eligibility criteria will be randomized in a 1:1 ratio to either real neurofeedback or sham feedback, with identical visit structure and procedures across groups.

The intervention will use an online neurofeedback pipeline to estimate right DLPFC activation from fNIRS signals in real time and present a visual activation bar to guide volitional downregulation of the target region during slow-wave acoustic cueing. The sham condition will use the same interface, cueing, and workflow but with feedback parameters configured to substantially weaken effective coupling between the displayed feedback and the participant's instantaneous neural state. fNIRS will be recorded across all training sessions, and ECG will be recorded during the first formal training session only to quantify heart rate and heart rate variability and to support mechanistic analyses of short-term brain-heart coupling during the task.

Clinical outcomes will focus on changes in anxiety severity over time, assessed at baseline, at the end of treatment, and at 3-month follow-up. Neurophysiological endpoints will be derived from the first formal session to characterize task-related right DLPFC downregulation, interhemispheric DLPFC synchrony, and cardiac autonomic responses during the neurofeedback task. Safety and tolerability will be evaluated by comparing the incidence and profile of adverse events between groups throughout the intervention period. In addition, both groups will receive matched, guideline-informed cognitive-behavioural therapy (CBT) during the intervention period as background standard care, and any clinically indicated psychotropic medication use during follow-up will be documented for analytic control.

ELIGIBILITY:
Inclusion Criteria:

* (i) Women aged 18-45 years, right-handed;
* (ii) Diagnosis of recurrent pregnancy loss (RPL), defined as ≥2 consecutive spontaneous pregnancy losses occurring before 28 weeks of gestation;
* (iii) Not currently pregnant, or currently in a missed miscarriage state;
* (iv) Meet DSM-5 diagnostic criteria for an anxiety disorder, with at least moderate severity, defined as Clinical Global Impression-Severity (CGI-S) ≥4;
* (v) Hamilton Anxiety Rating Scale (HAMA) ≥16, with 17-item Hamilton Depression Rating Scale (HAMD-17) <17, to ensure anxiety is the predominant affective disturbance.

Exclusion Criteria:

* (i) Markedly unstable blood pressure (systolic BP >180 mmHg or <90 mmHg);
* (ii) Clinically important comorbid organic diseases, including but not limited to hyperthyroidism, history of atrial fibrillation, sinus bradycardia, major neurological disorders, cerebrovascular disease, or severe pulmonary disease;
* (iii) Significant suicide risk, judged by psychiatric assessment to be unsuitable for study participation;
* (iv) Other severe psychiatric disorders, including substance use disorder, schizophrenia, delusional disorder, unspecified psychotic disorder, bipolar disorder, or delirium;
* (v) Use of any oral antidepressant, anxiolytic, or antipsychotic medication within the past 4 weeks, or fluoxetine within the past 6 weeks, or any long-acting injectable antipsychotic within the past 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
the between-group difference in treatment response | Day 0 (baseline, pre-intervention); Day 24 (end of treatment, within 1 hour after completion of training); 3 months after Day 24.
  The investigators will compare the overall proportion of participants achieving response in the real neurofeedback group versus the sham-feedback group across the post-treatment follow-up period, defined by two timepoints: end of treatment and 3-month follow-up. Anxiety symptoms will be assessed using the Hamilton Anxiety Rating Scale (HAMA; ; 14 items, each scored 0-4; total score range 0-56; higher scores indicate greater anxiety severity), and treatment response will be defined a priori as a reduction of at least 50% in total HAMA score from baseline.

SECONDARY OUTCOMES:
Between-group difference in remission rate. | Day 0 (baseline, pre-intervention); Day 24 (end of treatment, within 1 hour after completion of training); 3 months after Day 24.
  Remission will be defined as HAMA total score less than 8 together with a Clinical Global Impression-Improvement (CGI-I) score of 1 (very much improved) or 2 (much improved).
Between-group difference in continuous HAMA scores. | Day 0 (baseline, pre-intervention); Day 24 (end of treatment, within 1 hour after completion of training); 3 months after Day 24.
  Anxiety severity will be measured using the Hamilton Anxiety Rating Scale (HAMA; 14 items, each scored 0-4; total score range 0-56; higher scores indicate greater anxiety severity). HAMA total score will be analysed as a continuous outcome to evaluate group, time, and group-by-time effects.
Between-group difference in downregulation of right DLPFC HbO activation. | Day 4 after randomisation (first formal training day).
  During the slow-wave acoustic cueing-assisted neurofeedback task, fNIRS will be used to quantify participants ability to volitionally downregulate HbO activation in the right dorsolateral prefrontal cortex, and differences between groups will be compared.
Between-group difference in interhemispheric synchronisation within the DLPFC. | Day 4 after randomisation (first formal training day).
  During the slow-wave acoustic cueing-assisted neurofeedback task, wavelet transform coherence (WTC) will be used to estimate the time-frequency coherence distribution between homologous left and right DLPFC channels as an index of interhemispheric synchrony and functional coupling. WTC values will be Fisher z-transformed and averaged within the target frequency band 0.01-0.05 Hz and within the task-relevant time window to derive an individual-level synchronisation metric for between-group comparison.
Between-group difference in baseline-corrected heart-rate change. | Day 4 after randomisation (first formal training day).
  During the slow-wave acoustic cueing-assisted neurofeedback task, baseline-corrected changes in heart rate (HR) will be compared between groups to evaluate between-group differences in acute cardiac autonomic responses.
Between-group difference in HRV spectral power at 0.0167 Hz. | Day 4 after randomisation (first formal training day).
  Using wavelet-based time-frequency analysis, the investigators will compare between-group differences in HRV spectral power at 0.0167 Hz (corresponding to the 60-second cycle and within the very-low-frequency range of HRV) to characterise autonomic rhythmic responses to the neurofeedback task and slow-wave rhythmic cueing.
Between-group difference in adverse events during the intervention period. | From Day 1 (start of adaptation training) through Day 24 (end of treatment).
  Specifically, the investigators will compare the overall proportion of participants experiencing at least one adverse event (AE) in the real neurofeedback group versus the sham-feedback group, and will additionally compare the occurrence of prespecified AE categories, including but not limited to mild dizziness or somnolence, transient bradycardia- or blood-pressure-related discomfort, and headache or nausea.

OTHER OUTCOMES:
The indirect effect of group assignment (real neurofeedback vs sham feedback) on HR change through change in right DLPFC activation. | Day 4 after randomisation (first formal training day).
The indirect effect of group assignment on 3-month anxiety improvement through change in right DLPFC activation | Day 4 after randomisation (first formal training day) and 3 months after Day 24.
The indirect effect of group assignment on 3-month anxiety improvement through HR change | Day 4 after randomisation (first formal training day) and 3 months after Day 24.
Model performance metrics | Day 4 after randomisation (first formal training day).
  Operational performance of the online neurofeedback pipeline will be quantified, including mean per-frame total processing time (computation plus rendering) and frame-drop rate, as objective indicators of system stability and usability.
Blinding assessment. | 3 months after Day 24.
  A standardised questionnaire will be administered at 3-month follow-up to evaluate blinding integrity. Participants will rate their perceived group assignment using a 5-point scale (0-4): 0, certain not in the experimental group; 1, uncertain but leaning not experimental; 2, unable to judge; 3, likely in the experimental group; 4, very certain in the experimental group. Subsequent analyses will quantify blinding success and compare results between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Tao, MM, Principal Investigator — Shenyang Medical College; Yun-En Liu, MD, Study Chair — Shenyang Medical College; Fei Meng, MD, Study Director — Central Hospital Affiliated to Shenyang Medical Collage
Locations (1):
- Central Hospital Affiliated to Shenyang Medical Collage, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol